CLINICAL TRIAL: NCT00674908
Title: A Single Blind, Multicentric, Comparative, Vaccine Interchangeability Trial of Shan 5 (Liquid) and Easy Five (Liquid) [Diphtheria-Tetanus- Pertussis, Hepatitis B and Hib Pentavalent Combination Vaccines] in Indian Infants.
Brief Title: Phase IV Interchangeability Study of a Liquid Pentavalent Combination Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shantha Biotechnics Limited (Industry)
Responsible Party: Head Clinical Research and Medical Affairs, Shantha Biotechnics Limited
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SBL/DTPwHB-Hib/INT/2007/0200
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2009-06

CONDITIONS: Diphtheria; Tetanus; Pertussis; Hepatitis B; Haemophilus Influenzae Type B
Keywords: Vaccine; Prevention; Diphtheria; Tetanus; Pertussis; Hepatitis B; Haemophilus influenzae type b; Vaccine interchangeability; Single vs mixed sequence; Healthy infants
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Haemophilus Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shan 5 (Experimental): Diphtheria, tetanus, whole cell pertussis, recombinant hepatitis B and Hib tetanus toxoid conjugate pentavalent liquid combination vaccine
  Interventions: Biological: Shan 5
- Easy 5 (Active Comparator): Diphtheria, tetanus, whole cell pertussis, recombinant hepatitis B and Hib conjugate pentavalent liquid combination vaccine
  Interventions: Biological: Easy Five

INTERVENTIONS:
Biological: Shan 5 — Diphtheria, tetanus, whole cell pertussis, recombinant hepatitis B and Hib tetanus toxoid conjugate pentavalent liquid combination vaccine
  Arms: Shan 5
Biological: Easy Five — Diphtheria, tetanus, whole cell pertussis, recombinant hepatitis B and Hib conjugate pentavalent liquid combination vaccine
  Arms: Easy 5

SUMMARY:
The objective of this study is to compare the Safety and Immunogenicity of a mixed sequence of 2 different pentavalent vaccines (Diphtheria-Tetanus- Pertussis, Hepatitis B and Hib combination Vaccines) with single sequence of Shan 5 in infants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children in the age group six to eight weeks
* Born after a normal gestational period (36 - 42 weeks)
* Mother's HBsAg assured negative.
* Father, mother or legally acceptable representative properly informed about the study and having signed the informed consent form.
* Parents willing to fill the Diary Card

Exclusion Criteria:

* Administration of immunoglobulin or any blood products since birth.
* Use of any investigational, on-registered drug, or vaccine other than the study vaccine (with the exception of OPV & BCG vaccine) during the study period or within 30 days preceding the first dose of the study vaccine.
* Previous vaccination or evidence of infection with DTP or Hib.
* History of allergic disease or reaction likely to be exacerbated by any component of the vaccine including allergy to antibiotics.
* Major congenital or hereditary immunodeficiency.
* Infants having evidence of disease or fever, history of allergic disease or persistent hematological, hepatic, renal, cardiac or respiratory disease and signs of a CNS disorder at the time of vaccination.
* Infants showing any of the following reactions after any dose of study vaccine will be withdrawn for subsequent doses: body temperature more than 40.4 degree Celsius, persistent screaming or crying for 3 hours within 48 hours of vaccination, seizures, encephalopathy and hypersensitivity reaction.
* Parent/s or guardian of subject unable to maintain diary card
* Simultaneous participation in any other clinical study

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Seroprotection rates for Diphtheria, Tetanus, Pertussis, Hepatitis B and Hib following 3 doses of the vaccines in a single and mixed sequence regimen. | 4 months

SECONDARY OUTCOMES:
Solicited and unsolicited local and systemic adverse events following vaccination | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Raman Rao, MD, Study Director — Shantha Biotechnics Limited
Locations (3):
- India (3):
  - Smt NHL Municipal Medical College and LG Hospital, Ahmedabad, Gujarat
  - Kempegowda Institute of Medical Sciences, Bangalore, Karnataka
  - Deenanath Mangeshkar Hospital, Pune, Maharashtra